CLINICAL TRIAL: NCT06940037
Title: The Impact of Biological Mechanisms of Aging on Response Variability to Resistance Training in Older Adults (BRIO): A Randomized, Placebo-controlled Trial of Progressive Resistance Training in Older Adults.
Brief Title: The Impact of Biological Mechanisms of Aging on Response Variability to Resistance Training in Older Adults
Acronym: BRIO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Tufts University Jean Mayer USDA Human Nutrition Research Center on Aging (Other)
Responsible Party: Principal Investigator, Nathan K. LeBrasseur, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 24-010008; R01AG089150 (NIH)
Record Dates: First submitted 2025-01-16; First posted 2025-04-23 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-08

CONDITIONS: Aging; Mobility Disability
Keywords: aging; mobility; exercise; senescence; DNA methylation; skeletal muscle
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Progressive Resistance Training vs. Health Education
Who Masked: Investigator, Outcomes Assessor
Masking Description: Data analysis team
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Progressive Resistance Training (Other): participants will attend exercise session 3 times per week.
  Interventions: Other: Progressive Resistance Training
- Health Education (Other): participants will attend health educations classed 1 time per week.
  Interventions: Other: Health Education

INTERVENTIONS:
Other: Progressive Resistance Training — 3 times a week
  Arms: Progressive Resistance Training
Other: Health Education — once a week
  Arms: Health Education

SUMMARY:
To critically examine biological, clinical, and behavioral modulators of progressive resistance training-associated exercise response heterogeneity in physical function and whole-body metabolism in older adults.

ELIGIBILITY:
Inclusion Criteria:

* aged greater than or equal to 65 years
* sedentary (Community Healthy Activities Model Program for Seniors physical activity questionnaire to identify and exclude persons engaged in regular (125 min/week or more) moderate intensity physical activity
* at risk for mobility disability score of less than or equal to 10 (but greater than 3) on the SPPB
* willing to be randomized into HE or PRT
* willing to be transported or transport themselves to the clinical sites for the intervention and assessments

Exclusion Criteria:

* unwillingness to provide informed consent
* participation in lifestyle or pharmacologic intervention trial or structured program of exercise training in the past 6 months
* an SPPB score of less than or equal to 3
* osteoarthritis or condition with joint pain limiting daily life activities
* significant weight loss or gain (7.5% of body weight) in past six months
* current anti-coagulant or anti-platelet therapy (Coumadin, Eliquis, Pradaxa, Xarelto, heparin, Lovenox, Plavix)
* clinically significant abnormality in any of the screening laboratory values, including those identified as outside of the "normal limits', that are deemed to be of concern for participation in the study by the study physician
* acute or terminal illness
* Mini Mental State Exam (MMSE) <23
* myocardial infarction in the previous 6 months or other symptomatic coronary artery disease
* New York Heart Association Class III or IV congestive heart failure
* serious conduction disorder (e.g., 3rd degree heart block), uncontrolled arrhythmia, or new Q waves or ST-segment depressions (>3 mm) on ECG
* chronic obstructive pulmonary disease requiring oxygen therapy
* upper or lower extremity fracture in the previous 6 months
* uncontrolled hypertension (150/90 mm Hg)
* neuromuscular diseases and/or drugs which affect neuromuscular function
* current use of anabolic steroids, growth hormone, replacement androgen therapy, anti-androgen therapy
* allergy to lidocaine
* presence of significant liver or renal disease (eGFR < 45 mL/min)
* diagnosis of type I diabetes mellitus or insulin requiring type 2 diabetes mellitus
* HbA1c > 7%
* BMI <21 or >35 for men or >40 for women
* excessive alcohol intake (>14 alcoholic beverages per wk.)
* current tobacco use
* current participation in any interventional clinical trial
* current use of weight loss medications

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-08-11 (Actual); Primary Completion 2029-08-31 (Estimated); Study Completion 2030-08-31 (Estimated)

PRIMARY OUTCOMES:
Precisely define the variability in changes in physical function | baseline, 6 months
  Measured by the Short Physical Performance Battery (SPPB), a 0-12 categorical scale of walking speed, standing balance, and repeated sit-to-stand time, with higher scores reflecting better physical function.
Precisely define the variability in changes in blood glucose concentrations in response to a meal tolerance test | baseline, 6 months
  Blood glucose concentrations (millimoles/liter) will be measured in response to a physiologically relevant meal challenge. Lower values are indicative of better metabolic health.

SECONDARY OUTCOMES:
Precisely define the variability in changes in skeletal muscle size. | baseline, 6 months
  Measured by computed tomography scans of the mid-thigh. Larger muscle cross-sectional area (cm^2) reflects a greater quantity of skeletal muscle.
Precisely define the variability in changes in skeletal muscle strength. | baseline, 6 months
  Measured by the one-repetition maximum, in newtons, on a leg press device, with higher scores reflecting greater skeletal muscle strength.
Precisely define the variability in changes in six-minute walk distance. | baseline, 6 months
  Measured by the distance (meters) walked in six minutes, with longer distances reflecting better physical function.
Precisely define the variability in insulin secretion in response to a mixed meal tolerance test. | baseline, 6 months
  Blood insulin concentrations (pmol/L) will be measured in response to a physiologically relevant meal challenge. Insulin concentrations in a physiological range reflect better metabolic health, while low insulin concentrations can reflect an impaired insulin response and high insulin concentrations can reflect peripheral insulin resistance.
Precisely define the variability in changes in the percentage of glycated hemoglobin in the blood. | baseline, 6 months
  Measured by the percentage of glycated hemoglobin in the blood (often referred to as HbA1c). A lower percentage of HbAlc reflects lower blood glucose concentrations over the past two to three months.
Precisely define the variability in changes in blood lipids. | baseline, 6 months
  Blood lipids, including total cholesterol, low density lipoproteins (LDLs), high density lipoproteins (HDLs), and triglycerides will be measured. Lower levels of total cholesterol (mg/dL), LDLs (mg/dL), and triglycerides (mg/dL), and higher levels of HDLs (mg/dL), are reflective of better metabolic health.
Precisely define the variability in changes in waist-to-hip ratio. | baseline, 6 months
  The circumference (cm) of the waist and hips will be measured and a ratio will be calculated. A lower waist-to-hip ratio is reflective of a better body composition (less central obesity or visceral fat).

CONTACTS AND LOCATIONS:
Overall Officials: Nathan LeBrasseur, Ph.D, MS, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Jean Mayer USDA Human Nutrition Research Center on Aging, Tufts University, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No